CLINICAL TRIAL: NCT02100384
Title: Long Term Comparison of Ultrasonic and Hand Instrumentation in the Maintenance of Peri-implant Tissues: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2013:174
Record Dates: First submitted 2014-03-12; First posted 2014-03-31 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2015-10

CONDITIONS: Determination of Clinical Effects; Presence of Inflammatory Cytokines; Patients Perception of Discomfort; Titanium Scalers; Ultrasonics
Keywords: peri implant; Maintenance; Ultrasonic; Scalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasonics (Active Comparator): Ultrasonic instrumentation for peri-implant maintenance
  Interventions: Procedure: Peri-implant maintenance
- Scalers (Active Comparator): Titanium Scalers instrumentation for peri-implant maintenance
  Interventions: Procedure: Peri-implant maintenance

INTERVENTIONS:
Procedure: Peri-implant maintenance — The peri-implant maintenance will be performed by two experienced Registered Dental Hygienists with titanium scalers or ultrasonic instrumentation

SUMMARY:
Nowadays, dental implants are a very attractive and affordable treatment option for patients. According to the American Society of Implant Dentistry the dental implant market in the U.S is projected to reach $1.3 billion by 20101. Despite the high success rates of dental implants, it is clear that osseointegrated implants are susceptible to diseases. The prevalence of dental implant complications are rising as the number of individuals that are receiving implant treatment is also increasing. One of these peri-implant complications is an inflammatory condition known as peri-implant mucositis that occurs in 64.6% to 80% of the implant population.

The lack of preventive maintenance therapy in subjects with peri-implant mucositis is associated with a high incidence of peri-implantitis, which eventually may lead to implant loss. One important method in the prevention of peri-implant mucositis is the reduction in plaque accumulation, through individual oral hygiene procedures and regular peri-implant professional maintenance. It is highly important that patients be educated about the importance of developing good oral hygiene habits and to attend regular periodontal maintenance appointments. The clinicians have to recognize the significance of monitoring and maintaining peri-implant health.

Unfortunately, it is unclear which of the different maintenance regimens and treatments strategies for peri-implant mucositis and peri-implantitis are more effective. There is lack of information about which peri-implant maintenance protocol offers the best outcome in terms of reduction of inflammation and improved patient comfort. According to Grusovin et al, "there is only low quality evidence for which are the most effective interventions for maintaining or recovering health of peri-implant soft tissues and there is no reliable evidence as to which regimens are most effective for long term maintenance". Moreover, current approaches to implant maintenance are somewhat haphazard and not standardized.

It is assumed that what is appropriate for teeth is also beneficial for implants; as stated by Persson et al, 2010 "therapies proposed for the management of peri-implant diseases are currently based on the evidence available from the treatment of periodontitis". Two conventionally used methods of biofilm and calculus removal from teeth in North America are hand instruments (curettes and scalers) and ultrasonics. In teeth these two modalities of treatment have been studied extensively; conversely, there are fewer studies on dental implants. Renvert et al, 2008 concluded that mechanical non-surgical treatment might be effective to treat peri-implant mucositis but not peri-implantitis; however, the data supporting this literature review was scarce. The same research group compared ultrasonic instrumentation with specific-implant tips to titanium curettes in the treatment of peri-implantitis founding no group differences in the treatment outcomes with improvements in plaque and bleeding scores but no effects on probing depths. In addition, both methods failed to eliminate or reduce bacterial counts and no group differences were found in the ability to reduce the microbiota in a six months period.

One of the main concerns for dental implants is that metal scalers and ultrasonics generate a roughened surface on the implant, which in turn facilitates plaque accumulation and therefore makes maintenance of plaque free surfaces more difficult. It was observed in a recent study that special coated scalers and ultrasonic tips have been shown in vitro to be compatible with implant surfaces, however this has not been confirmed in vivo. The previous finding is in agreement with a current study, which demonstrated that the roughness values of the titanium surface of implants treated with piezoelectric ultrasonic scalers with a newly developed metallic tip and plastic hand curettes, are equal to the surface's roughness of untreated implants. Mann et al, 2012 showed in an in vitro study that plastic-coated scalers cause minimal damage to the implant surface but leave plastic deposits behind on the implant surface, suggesting further research is needed to evaluate the use of such plastic tips in the debridement of implants.

An additional factor, in evaluating the efficacy of different instrumentation in peri-implant maintenance, which needs to be taken into consideration, is patient perception. There is currently no data evaluating patient perception of comfort in regards to hand vs. ultrasonic instrumentation. This information is very important because should both methods of debridement be considered of equal efficacy, patient preference may play a role in the practitioner's selection of instrumentation. Knowing that patient comfort will increase the patient's compliance to the maintenance therapy, further evaluation of this factor is necessary.

DETAILED DESCRIPTION:
Long term comparison of ultrasonic and hand instrumentation in the maintenance of peri-implant tissues: A randomized clinical trial

Objective

The aim of this study is to determine the clinical effects, presence of inflammatory cytokines, and the patients' perceived discomfort by comparing titanium scalers to ultrasonic instrumentation using implant inserts in a patient population with healthy peri-implant tissues and implants with peri-implant mucositis during a one-year period of peri-implant maintenance.

Hypothesis

There are insufficient studies in the literature to guide the clinician which technique will offer better results in maintaining health or in decreasing inflammation long term around dental implants during peri-implant maintenance. It is postulated in this study that (1) peri-implant therapy will have a beneficial clinical effect, will decrease the presence of inflammatory cytokines and will be well tolerated by the patient population and that (2) there will be no differences in the outcomes between the two peri-implant maintenance therapies.

Materials and Methods

Previous approval by the Biomedical Research Ethics Board of the University of Manitoba a randomized clinical trial will be conducted between May, 2014 and May, 2015 at the Periodontics Clinic of the University of Manitoba. The Oral Biology Laboratory of the University of Manitoba will perform the analysis of samples of the peri-implant crevicular fluid. The Consolidated Standards of Reporting Trials, CONSORT Statement will be followed.

66 participants with at least one single dental implant will be recruited and randomly assigned to one of the two peri-implant maintenance groups. Subjects enrolled in the study will be regular patients of the Periodontics Graduated Clinic at the University of Manitoba, Faculty of Dentistry. Each participant will sign a written informed consent. The randomization will be computer-generated by a second person not involved in the study.

A total of 352 sites (6sites/implant) will be studied. Cohen effect size has been used to calculate the sample size. Small to medium effect size ranges by Cohen: 0.2mm to 0.5mm. In addition, independent t-test with alpha=0.05, power (1-beta) =80%, 95% confidence interval and two tailed test. Allocation ratio, n1/n2=1. G*Power 3.1.7 software was used in sample size calculation. An attrition rate of 6 participants was calculated.

A code will be assigned to each participant. Only the research coordinator will have access to the patients/codes matching list and its corresponding therapy. The peri-implant maintenance will be performed by two experienced Dental Hygienists previous intra and inter-examiner calibration. A single blinded calibrated examiner (MC) will do the recording of clinical findings and sampling at baseline, 3, 6 and 12 months.

The following are the inclusion criteria: (1) subjects having at least one single unit dental implant (2) probing depths no more than 5mm in 6 aspects around each implant (MB, B, DB, ML, L and DL), (3) no bone loss beyond 2mm/implant at baseline confirmed with periapical radiographs with a cone paralleling technique. The next criteria will be excluded from the study: (1) implant supported removable prostheses, (2) use of antibiotics within the preceding 3 months (3) smokers (4) missing exam at baseline.

The parameters to be assessed at 6 sites/implant are the following: (1) Modified plaque index by Mombelli (2) Modified gingival index by Mombelli, (3) probing depths (PD), (4) presence of keratinized gingiva (0, 0.5-1.5mm, 2 or greater), (5) recession (REC) distance between gingival margin and most occlusal point of restoration, (6) Cytokine levels in peri-implant crevicular fluid, 1 sample from the deepest site of implant(s) will be collected at baseline, 3, 6 and 12 months. In addition, patients will also be asked to fill in a pain questionnaire at the end of the study period (Visual analogue scale, VAS).

To collect the peri-implant crevicular fluid, the site will be isolated from saliva using cotton rolls and drying before the sampling. Periopaper strips (Oraflow) will be introduced at the deepest site of the implant sulcus for 30 sec. The volume of peri-implant crevicular fluid will be measured using a Periotron. Until further analysis strips will be store at -80C in sealed plastic tubes previously identified with a code corresponding to the name of the patient. Pro-inflammatory/pleiotropic cytokines, which are found during inflammatory processes at cellular level will be assess. The fluorescence based multiplex protein quantification system (BioPlex, BioRad, Hercules CA, USA) will be used to measure the following eight cytokines: GM-CSF, IFN-gamma, IL-2, IL-4, IL-6, IL-8, IL-10 and TNF-α.

Ethical Considerations

The patients will be asked to review and sign a written consent form. Only individuals involved in this study will have access to the data collected during the study. The records for each patient will be assigned with a unique number and will be stored by the principal investigator at her desk within the clinic premises. The master sheet linking the patient identifiers to the unique number will be stored in a safe in the clinic administrative office. In case of possible continuation of line of investigation, the data could be compared with new data (introduction of air abrasive). The master sheet and patient records will be shredded at the end of 4-5 years. To thank them for their participation in the study they will receive a free maintenance appointment at the end of the study (12 months).

Relevance of the study

This study is relevant because there is currently no long term in vivo studies that determine the effectiveness of peri-implant maintenance and also the possible differences and/or similar outcomes between curettes and ultrasonics in the peri-implant maintenance protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with healthy peri-implant tissues and implants with peri-implant mucositis

Exclusion Criteria:

* All others

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reduction of inflammation | 12 Months

SECONDARY OUTCOMES:
Probing depths | 0 - 3 - 6 - 9 and 12

OTHER OUTCOMES:
Cytokines | 12 Months
Patient comfort | 12 Months
Bleeding scores | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Castro, DDS, MSc, Principal Investigator — University of Manitoba; Anastassia Cholakis, DMD, Dip., Perio., FRCD(C), Study Director — University of Manitoba
Locations (1):
- University of Manitoba Faculty of Dentistry Periodontics Clinic, Winnipeg, Manitoba, Canada